CLINICAL TRIAL: NCT02631603
Title: Stop Exogenous Allergic Alveolitis (EAA) in Childhood: Healthy Into Adulthood - A Randomized, Double-blind, Placebo-controlled, Parallel-group Study to Evaluate Prednisolone Treatment and Course of Disease
Brief Title: Stop Exogenous Allergic Alveolitis (EAA) in Childhood
Acronym: chILD-EU_EAA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: After several years of recruitment only 4 patients were included. Study timelines for study completition too long. Decided to terminate trial.
Sponsor: Matthias Griese (Other)
Responsible Party: Sponsor-Investigator, Matthias Griese, Prof. Dr. med., Ludwig-Maximilians - University of Munich
Organization: Ludwig-Maximilians - University of Munich (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: StopEAA
Record Dates: First submitted 2015-11-29; First posted 2015-12-16 (Estimated); Results first posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Hypersensitivity Pneumonitis; Exogenous Allergic Alveolitis
Keywords: Children; Birds; Moulds
MeSH Terms: conditions — Alveolitis, Extrinsic Allergic | interventions — Prednisolone; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Experimental): Capsules of placebo will be taken for 3 months, same schedule as verum.
  Interventions: Drug: Placebo
- Prednisolone (Active Comparator): Oral prednisolone, anticipated dose:
  first month 0.5 mg/kg bw/d, second month 0.25 mg/kg bw/d, and third month 0.125 mg/kg bw/d in a single morning dose.
  Individual capsules will be prepared using rounded dose.
  Interventions: Drug: Prednisolone

INTERVENTIONS:
Drug: Placebo — Administer Placebo as anti-inflammatory
  Other Names: no other name
  Arms: Placebo
Drug: Prednisolone — Administer Prednisolone as anti-inflammatory
  Other Names: Decortin H
  Arms: Prednisolone

SUMMARY:
Stop exogenous allergic alveolitis (EAA) or hypersensitivity pneumonitis in childhood: healthy into adulthood - a randomized, double-blind, placebo-controlled, parallel-group study to evaluate prednisolone treatment and course of disease.

The hypothesis of the study is that the treatment with placebo will not be inferior in terms of Forced Vital Capacity (FVC) improvement than treatment with systemic steroids after 6 months treatment.

DETAILED DESCRIPTION:
After an initial steroid pulse given to all patients, patients will be allocated to the two treatments, i.e., oral prednisolone and Placebo.

Experimental intervention: Placebo Control intervention: Prednisolone Duration of intervention per patient: 3 months Follow-up per patient: 3 months

Primary Objective:

To evaluate outcome of EAA at 6 months and compare the medium term treatment with systemic steroids or placebo.

Secondary Objectives:

To evaluate the completeness and knowledge of standardized and pedantic allergen elimination in families with a child with EAA.

To evaluate the treatment of EAA with systemic steroids compared to placebo at 3 months.

To evaluate the safety of the treatment of EAA with outpatient usage of systemic steroids compared to Placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Newly or previously diagnosed but not appropriately treated EAA in children, adolescents and young adults, aged between 3 and 25 years. The diagnosis of EAA must be confirmed by independent review of the findings by an expert panel and must be based on the presence of at least 4 of the following findings:

   * History of appropriate allergen exposure
   * Restrictive lung function (FVC < 80% predicted for age and FVC/FEV1 < 1) testing, if appropriate for age (usually > 5 y)
   * Positive serum precipitins for bird/fungus exposed to (other allergens have rarely, if every been demonstrated in children)
   * Lymphocytosis in BAL (> 20% of cells are lymphocytes)
   * HRCT showing the characteristic nodular, linear or reticular opacities, and ground glass pattern with increased attenuation.
   * Lung biopsy demonstrating lymphocytic alveolitis, bronchiolitis, and non-caseating histiocytic granulomatas.
   * Controlled allergen exposure followed by characteristic reaction, including fever, coughing, restriction on lung function, hypoxemia/desaturation at rest or with exercise
2. Unchanged inhaled steroids if on; if off, no plans to introduce them in the following 6 months
3. Agreement to home visit by independent study physician

Exclusion Criteria:

1. Contraindication for usage systemic steroids
2. Critically ill patients needing respiratory support
3. Non-compliance with medical treatments and interventions
4. Women with childbearing potential and not practicing a medically accepted contraception during the trial and a positive pregnancy test (serum or urine) before and at the end of the trial. Reliable contraception are systematic contraceptives (oral, implant, injection) and diaphragm or condoms with spermicide.
5. Pregnancy and lactation.
6. Participation in another trial for EAA during the last 4 weeks or not beyond the time of 4 half-lives of the medication used. In the unlikely event a subject is already in another clinical study but not for EAA, that study must be stopped and the subject may be treated according to this protocol; a latency time between the two studies does not appear reasonable, as acute intervention is necessary for EAA. Treatment may be best done in the frame work of this protocol.

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-07-11 (Actual); Study Completion 2020-06-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Griese, Prof., MD, Study Director — Pediatric Pneumology, Ludwig-Maximilians-University Munich; Meike Hengst, MD, Principal Investigator — Pediatric Pneumology, Ludwig-Maximilians University Munich
Locations (7):
- Germany (7):
  - Klinikum der Universität München, Haunersches Kinderspital, München, Bavaria
  - Universitätsklinikum Frankfurt, Pneumologie, Allergologie, Mukoviszidose, Frankfurt am Main, Hesse
  - Justus-Liebig-Universität, Allgemeine Pädiatrie u. Neonatologie, Giessen, Hesse
  - Medizinische Hochschule Hannover, Hanover, Lower Saxony
  - Klinik für Kinder- und Jugendmedizin der Ruhr-Universität Bochum im St. Josef-Hospital, Bochum, North Rhine-Westphalia
  - Uniklinikum Essen, Pädiatrische Pneumologie, Essen, North Rhine-Westphalia
  - Klinik u. Poliklinik für Kinder- u. Jugendmedizin der Universität Leipzig, Leipzig, Saxony

IPD SHARING:
Plan to Share IPD: No
Equivalent to product information sheet

REFERENCES:
- [Result] Griese M, Stehling F, Schwerk N, Rosewich M, Jerkic PS, Rock H, Ruckes C, Kronfeld K, Sebah D, Wetzke M, Seidl E. Hypersensitivity pneumonitis: Lessons from a randomized controlled trial in children. Pediatr Pulmonol. 2021 Aug;56(8):2627-2633. doi: 10.1002/ppul.25513. Epub 2021 May 28. PMID 34048641

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Originally, it was planned to screen 60 subjects to include approximately 40 patients. From January 2015 to July 2016 due to difficulties in funding only 4 children were included in the trial. All met inclusion criteria, were randomized, and completed the trial.
Groups:
- Placebo: Capsules of placebo will be taken for 3 months.
  Placebo: Administer Placebo as anti-inflammatory
- Prednisolone: Oral prednisolone, anticipated dose:
  first month 0.5 mg/kg bw/d, second month 0.25 mg/kg bw/d, and third month 0.125 mg/kg bw/d in a single morning dose.
  Individual capsules will be prepared using rounded dose.
  Prednisolone: Administer Prednisolone as anti-inflammatory
Period: Overall Study
Arm/Group | Placebo | Prednisolone
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Prednisolone 1; Prednisolone 2; Prednisolone 3: Oral prednisolone, anticipated dose:
  first month after steroid pulse 0.5 mg/kg bw/d, second month 0.25 mg/kg bw/d, and third month 0.125 mg/kg bw/d in a single morning dose.
- Placebo: Capsules of placebo will be taken for 3 months.
- Total: Total of all reporting groups
Arm/Group | Prednisolone 1 | Placebo | Prednisolone 2 | Prednisolone 3 | Total
Number analyzed (Participants) | 1 | 1 | 1 | 1 | 4
Age, Customized [Number; unit: years] — Patients between 3 to 18 years
  years | 8.4 | 6.6 | 10.6 | 12.9 | 9.6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1 | 0 | 2
  Male | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 1 | 1 | 1 | 1 | 4
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 1 | 1 | 1 | 1 | 4
O2 saturation at rest [Number; unit: %] | 90 | 98 | 100 | 97 | 96.3

OUTCOME MEASURES:

1. Primary Outcome: Forced Vital Capacity (FVC).
Description: The relative change from baseline through month 6 compared to change from placebo of FVC.
Time Frame: 6 months
Measure: Number; unit: % predicted
Groups:
- Prednisolone 1; Prednisolone 2; Prednisolone 3: Oral prednisolone, anticipated dose:
  first month 0.5 mg/kg bw/d, second month 0.25 mg/kg bw/d, and third month 0.125 mg/kg bw/d in a single morning dose.
Arm/Group | Prednisolone 1 | Placebo | Prednisolone 2 | Prednisolone 3
Number analyzed (Participants) | 1 | 1 | 1 | 1
% predicted | 126 | 103 | 84 | 65

2. Secondary Outcome: Forced Vital Capacity (FVC)
Description: FVC measured in accordance to standarized protocol.
Time Frame: 3 months
Measure: Number; unit: % predicted
Arm/Group | Prednisolone 1 | Placebo | Prednisolone 2 | Prednisolone 3
Number analyzed (Participants) | 1 | 1 | 1 | 1
% predicted | 114 | 95 | 85 | 76

ADVERSE EVENTS:
Time Frame: 6 months
Description: The adverse events were collected during the study visits or during the telephone visits.
Arm/Group | Placebo | Prednisolone
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 3/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1) | Prednisolone (N=3)
Fever, headache, haematome, tiredness, hypertension (General disorders) | 1 (2) | 2 (3) — Besides the occurance of adverse events and their frequency also the affected organ system was collected in the study data.
Conjunctivitis (Eye disorders) | 1 (1) | 1 (1) — Besides the occurance of adverse events and their frequency also the affected organ system was collected in the study data.
Respiratory tract infection, candidiasis (Infections and infestations) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cushing habitus, hair growth, weight gain (Endocrine disorders) | 1 (1) | 1 (2)

LIMITATIONS AND CAVEATS:
The major limitation of this trial was its premature closure and the small number of patients included. This was due to several reasons: the study design was developed as work package within a limited research project. The anticipated enrolment was lower than expected. There was a lack of resources to carry on the clinical trial for the many years in view of the much lower incidences of this rare conditions than calculated before on available data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2014-12-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT02631603/Prot_000.pdf